CLINICAL TRIAL: NCT00977444
Title: Evaluation of a New Formulation Useful for the Osteoarthrosis Treatment
Acronym: EFO
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nucitec (Industry)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Sandra Garcia, Cindetec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEE-002-2007
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Osteoarthritis
Keywords: knee; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- kondrium (Experimental): intraarticular injections once month
  Interventions: Drug: kondrium
- kondrium f (Experimental)
  Interventions: Drug: kondrium f
- corticosteroid (Active Comparator): intraarticular injections once month
  Interventions: Drug: methyl prednisolone (corticosteroid)

INTERVENTIONS:
Drug: kondrium — intraarticular injections once month
  Arms: kondrium
Drug: kondrium f — intraarticular injections once month
  Arms: kondrium f
Drug: methyl prednisolone (corticosteroid) — intraarticular injections once month
  Other Names: corticosteroid
  Arms: corticosteroid

SUMMARY:
Abstract

Kondrium, is a pharmaceutical composition for the treatment of osteoarthritis (OA). This study was designed to evaluate the efficacy and safety of kondrium in the treatment of OA of knee.

A 3 month, randomized, double-blind, active-controlled, parallel-group study will be carried out. 117 patients with OA of the knee will be randomized to receive 1 intra-articular monthly injection of 5 mL of one of the following: 75 mg/mL of Kondrium, 82.5 mg/mL of Kondriumf or 8 mg/mL of methylprednisolone once a month during 3 months. The primary efficacy variable will be the change from baseline to final assessment in the Western Ontario and McMaster University OA index (WOMAC subscale score for pain), and Lequesne´s functional index.

DETAILED DESCRIPTION:
The WOMAC osteoarthritis index is a validated, multidimensional, disease specific, health status measure. It probes clinically important patient relevant symptoms in the areas of pain, stiffness and physical function in patients with hip and/or knee osteoarthritis. It consists of 24 questions in three separated subscales (5 questions on pain subscale, 17 questions on physical function subscales and 2 questions on stiffness subscale), each scored in analog scale from 0 to 10 points (0 representing no pain, 10 representing extreme pain). Each subscale score was weighed 10 points, thus 30 was the maximum punctuation for WOMAC total score.

The Lequesne index is a 10-question interview-style survey given to patients with osteoarthritis of the knee. It has 5 questions pertaining to pain or discomfort, 1 question dealing with maximum distance walked, and 4 questions about daily activities. The total questionnaire is scored on a 0 to 24 scale, with lower scores meaning less functional impairment.

ELIGIBILITY:
Inclusion Criteria:

* age > 40 years
* symptomatic evidence of OA in the knee for at least 1 year
* radiographic evidence of Kellgren and Lawrence grade II to IV OA of the knee
* no intra-articular injection of corticosteroids within the last 3 months

Exclusion Criteria:

* any history of adverse reaction to the study drugs
* current pregnancy status
* uncontrolled hypertension
* active infection
* undergone surgery/arthroscopy within three months
* diagnosis of radiographic OA of Kellgren and Lawrence grade I

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy variable is the change from baseline to final assessment in the Western Ontario and McMastern University OA index (WOMAC), and Lequesne´s functional index. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Amador, PhD, Principal Investigator — Hospital San Jose
Locations (1):
- Hospital San Jose, Querétaro City, Querétaro, Mexico

REFERENCES:
- [Derived] Caamano MDC, Garcia-Padilla S, Duarte-Vazquez MA, Gonzalez-Romero KE, Rosado JL. A Double-Blind, Active-Controlled Clinical Trial of Sodium Bicarbonate and Calcium Gluconate in the Treatment of Bilateral Osteoarthritis of the Knee. Clin Med Insights Arthritis Musculoskelet Disord. 2017 Feb 16;10:1179544116688899. doi: 10.1177/1179544116688899. eCollection 2017. PMID 28469486
- [Derived] Garcia-Padilla S, Duarte-Vazquez MA, Gonzalez-Romero KE, Caamano Mdel C, Rosado JL. Effectiveness of intra-articular injections of sodium bicarbonate and calcium gluconate in the treatment of osteoarthritis of the knee: a randomized double-blind clinical trial. BMC Musculoskelet Disord. 2015 May 13;16:114. doi: 10.1186/s12891-015-0568-4. PMID 25963758